CLINICAL TRIAL: NCT03460912
Title: Comparison of Different Types of Electrostimulation Probes for Intraoperative Nerve Monitoring During Thyroidectomy
Brief Title: Different Types of Electrostimulation Probes During IONM
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ozer Makay, Associate Professor Ozer Makay, Ege University
Other Study IDs: yturk1
Record Dates: First submitted 2018-02-05; First posted 2018-03-09 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Thyroid Diseases
Keywords: IONM; thyroidectomy; bipolar probe; monopolar probe
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants
  Interventions: Device: Bipolar and monopolar probes (SPESS MEDICA S.r.l. Via Buccari 16153 Genova (GE), Italy) administered to all participants.

INTERVENTIONS:
Device: Bipolar and monopolar probes (SPESS MEDICA S.r.l. Via Buccari 16153 Genova (GE), Italy) administered to all participants. — Bipolar and monopolar probes (SPESS MEDICA S.r.l. Via Buccari 16153 Genova (GE), Italy) administered to all participants.They compared each others(bipolar vs monopolar) via amplitudes and latency values.

SUMMARY:
Intraoperative nerve monitoring is often used in many centers during thyroidectomy. According to the investigators' knowledge, there's no study showing superiority between bipolar and monopolar stimulation probes used for nerve monitoring during thyroid surgery. In this study, the investigators aimed to compare two different types of probes and find out superiorities.Twenty-one patients who underwent primary total thyroidectomy or hemithyroidectomy were included in the study. During surgery, amplitude and latency values obtained in the same patient with both bipolar and monopolar stimulation probes from 10 different anatomical spots [vagal nerve, recurrent laryngeal nerve inferior portion, recurrent laryngeal nerve superior portion, external branch of superior laryngeal nerve (EBSLN)] were recorded prospectively, both when sheath was intact and after being dissected.

ELIGIBILITY:
Inclusion Criteria:

* who underwent thyroid surgery

Exclusion Criteria:

* Perioperative loss of electromyographic(EMG) signal (LOS) during intraoperative nerve monitorization
* patients with additional pathology that may affect vocal cord function,
* abnormal preoperative laryngeal examination
* history of thyroid, vocal cord or other neck surgery
* advanced cancer, RLN, esophageal or trachea invasion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consequtive patients who underwent thyroid surgery
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-06-26 (Actual); Primary Completion 2016-12-26 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Comparison of amplitude values of bipolar vs. monopolar stimulation | One week
  Bipolar and monopolar probes were compared regarding amplitudes(mA), at each spot and on both sides (right & left) via Wilcoxon Signed Rank Test.
Comparison of Latency values of bipolar vs. monopolar stimulation | One week
  Bipolar and monopolar probes were compared regarding latencies(ms) , at each spot and on both sides (right & left) via Wilcoxon Signed Rank Test.

SECONDARY OUTCOMES:
Comparison of stimulation with vs. without overlying fascia on nerve | One week
  The assessment was based on the presence or absence of nerve sheaths in this group in amplitude values via Wilcoxon Signed Rank Test.
Comparison of stimulation pre- vs. post-resection without overlying fascia on nerve | One week
  The assessment in this group was made according to pre- and post-resection amplitude values from vagus and recurrent nerve, that were compared to each other on both sides (right & left) and with both (bipolar & monopolar) probes via Wilcoxon Signed Rank Test.
Comparison of stimulation of inferior vs. superior parts of recurrent nerve. | One week
  The assessment in this group was based on the latency values between the inferior and superior part of the recurrent nerve via Wilcoxon Signed Rank Test.